CLINICAL TRIAL: NCT04793581
Title: Assessment of the Utility of the Pantheris SV System
Brief Title: Assessment of the Utility of the Pantheris Small Vessel (SV) System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Avinger, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMAGE BTK
Record Dates: First submitted 2021-01-29; First posted 2021-03-11 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral artery disease (PAD) below-the-knee atherectomy
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Atherectomy

STUDY DESIGN:
Intervention Model Description: Single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Other): Single-arm study
  Interventions: Device: Atherectomy

INTERVENTIONS:
Device: Atherectomy — Directional atherectomy of lesions below the knee.

SUMMARY:
A single-arm study to assess the utility of the Pantheris SV catheter in addressing peripheral artery disease in arteries located below the knee. Data will be collected on the percent stenosis pre- and post-atherectomy and then symptoms and adverse events noted at 30 days, 6 months, and 1 year after the procedure.

DETAILED DESCRIPTION:
This is a post-market, single-arm study of the optical coherence tomography (OCT)-guided directional atherectomy catheter, Pantheris SV. Patients presenting with reduced blood flow in the lower extremity arteries will under directional atherectomy, followed by adjunctive therapy as deemed necessary by the physician, and then adverse events and symptom resolution will be documented at 30 days, 6 months, and 1 year after the procedure. Primary safety endpoints are related to adverse events and will be assessed at the time of the procedure and at 30 days after the procedure. Effectiveness endpoints center on restoration of blood flow.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Target lesion in the infragenicular segment
* At least 1 pedal vessel noted in the foot
* Rutherford classification 3 to 6
* Willing to give informed consent

Exclusion Criteria:

* if female, is pregnant or breast feeding
* has had surgery or endovascular procedure within 30 days prior to the index procedure
* has planned surgery within 30 days after the index procedure
* had a major bleeding event within 60 days prior to the index procedure
* currently in the treatment phase of a drug or device trial
* has anticipated life span of less than 1.5 years
* is unwilling to present to the investigator at 30 days, 6 moths, or 1 year after the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Events | from procedure to 30 days post-procedure
  freedom from cardiovascular-related events
Technical success | At 1 day post-procedure
  defined as residual stenosis < 50 percent after atherectomy

SECONDARY OUTCOMES:
Procedure success | At 1 day post-procedure
  defined as residual stenosis < 30 percent post adjunctive therapy
Freedom from target vessel revascularization (TVR) | At 6 and 12 months post-procedure
  revascularization needed further
Primary patency | At 6 and 12 months post-procedure
  change in peak systolic velocity ratio (PSVR)
Ankle-Brachial Index (ABI) | At 6 and 12 months post-procedure
  change since index procedure
Rutherford Classificaiton | At 30 days, 6 months, and 1 year post-procedure
  Change since index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jaafer Golzar, MD, Study Chair — Avinger, Inc.
Locations (2):
- United States (2):
  - Advanced Cardiac and Vascular Centers, Grand Rapids, Michigan
  - Eastlake Cardiovascular PC, Saint Clair Shores, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khalili H, Jeon-Slaughter H, Armstrong EJ, Baskar A, Tejani I, Shammas NW, Prasad A, Abu-Fadel M, Brilakis ES, Banerjee S. Atherectomy in below-the-knee endovascular interventions: One-year outcomes from the XLPAD registry. Catheter Cardiovasc Interv. 2019 Feb 15;93(3):488-493. doi: 10.1002/ccd.27897. Epub 2018 Nov 30. PMID 30499198
- [Result] Schwindt AG, Bennett JG Jr, Crowder WH, Dohad S, Janzer SF, George JC, Tedder B, Davis TP, Cawich IM, Gammon RS, Muck PE, Pigott JP, Dishmon DA, Lopez LA, Golzar JA, Chamberlin JR, Moulton MJ, Zakir RM, Kaki AK, Fishbein GJ, McDaniel HB, Hezi-Yamit A, Simpson JB, Desai A. Lower Extremity Revascularization Using Optical Coherence Tomography-Guided Directional Atherectomy: Final Results of the EValuatIon of the PantheriS OptIcal COherence Tomography ImagiNg Atherectomy System for Use in the Peripheral Vasculature (VISION) Study. J Endovasc Ther. 2017 Jun;24(3):355-366. doi: 10.1177/1526602817701720. Epub 2017 Apr 10. PMID 28393673